CLINICAL TRIAL: NCT05180474
Title: First-in-human, Open-label, Dose-escalation Trial With Expansion Cohorts to Evaluate Safety of GEN1047 in Subjects With Malignant Solid Tumors
Brief Title: GEN1047 for Solid Tumors - First in Human (FIH) Trial
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1047-01; NL82658.056.23 (Registry Identifier: CCMO (The Netherlands)); 1007620 (Registry Identifier: Research Summaries Database (UK)); 2021-001790-23 (EudraCT Number); 2024-510722-10 (Other: EU Trial (CTIS) Number); RECF-004736 (Other: The French National Cancer Institute)
Record Dates: First submitted 2021-11-08; First posted 2022-01-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer, Breast Neoplasms; Endometrial Cancer, Endometrial Neoplasm; Ovarian Cancer, Ovarian Neoplasms; Squamous Non Small Cell Lung Cancer (NSCLC-SCC)
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GEN1047 (Experimental)
  Interventions: Biological: GEN1047 is a bispecific antibody that induces T-cell mediated cytotoxicity of B7H4-positive tumor cells.

INTERVENTIONS:
Biological: GEN1047 is a bispecific antibody that induces T-cell mediated cytotoxicity of B7H4-positive tumor cells. — GEN1047 will be administered as an intravenous infusion. The dose-levels will be determined by the starting dose and the escalation steps taken in the trial.
  Other Names: DuoBody®-CD3-H101GxB7H4

SUMMARY:
The purpose of this trial is to measure the following in participants with solid tumors who receive GEN1047:

* The side effects seen with GEN1047
* What the body does with GEN1047 once it is administered
* What GEN1047 does to the body once it is administered
* How well GEN1047 works against solid tumors

The estimated trial duration for an individual participant is 8 months, consisting of a 28-day screening period, an estimated 3 month treatment period (the duration of treatment may vary for each participant), and an estimated 4 month post-treatment follow-up period (the duration of follow-up may vary for each participant). All participants will receive active drug; no one will be given placebo.

DETAILED DESCRIPTION:
The trial is an open-label, multi-center safety trial of GEN1047. The trial consists of two parts: a dose escalation part ("escalation" - phase 1) and an expansion part ("expansion" - phase 2a). The goal of the dose escalation part is to find out if GEN1047 is safe in participants with specific solid tumors and to find the best dose(s). In the expansion part of the trial up to two doses of GEN1047 will be tested.

ELIGIBILITY:
Key Inclusion Criteria:

Criteria - Escalation Part:

* Participant must have histologically or cytologically confirmed solid tumor(s) in any of the following selected indications for which there is no further available standard therapy likely to confer clinical benefit (or participant is not a candidate or has previously refused such earlier available therapy), and for whom, in the opinion of the investigator, experimental therapy with GEN1047 may be beneficial (breast cancer, endometrial cancer, ovarian cancer, NSCLC-SCC.
* Participants with ovarian cancer must have documented progressive disease (PD) on or after last prior treatment and within 60 days of screening.
* Must be at least 18 years of age (or the legal age of consent in the jurisdiction in which the trial is taking place) on the day of signing informed consent.
* Must have either recurrence after, or progression on or lack of response to available relevant standard of care (SoC) anticancer therapies; or are deemed intolerant to or ineligible for, standard curative therapy in the recurrent setting.
* Must have at least 1 measurable lesion per RECIST v1.1. The measurable lesion(s) must be outside the field of radiation therapy (RT) if there was prior treatment with RT.
* Must have an Eastern Cooperative Oncology Group performance status (ECOGPS) score of 0 to 1 at Screening and on C1D1 pretreatment.
* Should provide a tumor tissue sample during the Screening period and prior to C1D1.
* Provide all tumor-assessing pre-trial CT scans since failure of last prior therapy.

Criteria - Expansion Part Stage 1, 1b and Stage 2:

* Participants must have documented PD according to RECIST v1.1 on or after last prior treatment with latest scan performed a maximum of 28 days prior to the first dose.
* Participant must have advanced (unresectable) or metastatic, histologically confirmed diagnosis (breast cancer, endometrial cancer, ovarian cancer.
* Must be a female and at least 18 years of age (or the legal age of consent in the jurisdiction in which the trial is taking place) at the time of consent.
* Must have at least 1 measurable lesion per RECIST v1.1 as assessed by local investigator.
* Must have an ECOG- PS score of 0 to 1 at Screening and on Cycle 1 Day 1 (C1D1) pretreatment.
* Must submit a tumor tissue sample during the Screening period and prior to C1D1.
* Provide all tumor-assessing pre-trial CT scans since failure of last prior therapy.

Key Exclusion Criteria:

* Significant cardiovascular impairment within 6 months of the first dose of trial drug.
* Participant with new or progressive brain metastases or spinal cord compression.
* Participant has been exposed to any prior therapy with a compound targeting CD3 and/or B7H4 or cell based therapies.
* Current pneumonitis (any grade) including any radiological change of ongoing pneumonitis at baseline or history of non-infectious drug-, immune-, or radiation-related pneumonitis that required steroid.

Note: Other protocol defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Escalation: Number of Participants with Dose Limiting Toxicities (DLT) | From the first Cycle (Cycle length=21 days) in each cohort
  DLTs will be graded for severity according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), v5.0.
Escalation: Number of Participants with Treatment Emergent Adverse Events (TEAEs) | From first dose date up to end of the safety follow up period, 30 days after last dose (approximately 4 months)
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAE is defined as an AE occurring or worsening between the first dose of study drug and 30 days after the last dose received.
Expansion: Objective Response Rate (ORR) | Up to 5 years
  ORR is defined as percentage of participants with best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) based on RECIST v1.1.

SECONDARY OUTCOMES:
Escalation and Expansion: Clearance | Predose and postdose at multiple timepoints of each Cycle (Cycle length=21 days)
Escalation and Expansion: Volume of Distribution (Vd) | Predose and postdose at multiple timepoints of each Cycle (Cycle length=21 days)
Escalation and Expansion: Area Under the Concentration-time Curve from Time 0 to Time of Last Dose (AUClast) | Predose and postdose at multiple timepoints of each Cycle (Cycle length=21 days)
Escalation and Expansion: AUC From Time Zero to Infinity (AUC0-inf) | Predose and postdose at multiple timepoints of each Cycle (Cycle length=21 days)
Escalation and Expansion: Maximum (Peak) Plasma Concentration (Cmax) | Predose and postdose at multiple timepoints of each Cycle (Cycle length=21 days)
Escalation and Expansion: Time to Reach Cmax (Tmax) | Predose and postdose at multiple timepoints of each Cycle (Cycle length=21 days)
Escalation and Expansion: Plasma Trough (Pre-dose) Concentrations (Ctrough) | Predose and postdose at multiple timepoints of each Cycle (Cycle length=21 days)
Escalation and Expansion: Elimination half-life (t 1/2) | Predose and postdose at multiple timepoints of each Cycle (Cycle length=21 days)
Escalation and Expansion: Number of Participants with Anti-Drug Antibody (ADA) | Up to 5 years
Escalation: ORR | Up to 5 years
  ORR is defined as percentage of participants with BOR of confirmed CR or confirmed PR based on RECIST v1.1.
Escalation and Expansion: Duration of Response (DOR) | Up to 5 years
  DOR is defined as the time from the first documented response to the first documented progression or death due to any cause.
Escalation and Expansion: Time to response (TTR) | Up to 5 years
  Time to response (TTR) is defined as the time from the date of Cycle 1 Day 1 (C1D1) to the first documented response of either confirmed CR or confirmed PR.
Escalation and Expansion: Disease control rate (DCR) | Up to 5 years
  The disease control rate (DCR) is defined as the percentage of participants with BOR of confirmed CR, confirmed PR, or stable disease (SD) according to RECIST v1.1
Expansion: Progression Free Survival (PFS) | Up to 5 years
  PFS is defined as the time from the date of C1D1 to the date of the first documented progression or death due to any cause, whichever occurs earlier according to RECIST v1.1.
Expansion: Overall Survival (OS) | Up to 5 years
  OS is defined as the time from date of C1D1 to date of death due to any cause.
Expansion: Number of Participants with TEAEs | From first dose date up to end of the safety follow up period, 60 days after last dose (approximately 5 months)
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAE is defined as an AE occurring or worsening between the first dose of study drug and 30 days after the last dose received.

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (36):
- United States (6):
  - UCLA Department of Medicine Hematology Oncology, Los Angeles, California
  - Yale University - Yale Cancer Center, New Haven, Connecticut
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Case Western Reserve University, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Belgium (2):
  - Antwerp University Hospital, Edegem
  - Universitair Ziekenhuis Leuven, Leuven
- Rigshospitalet (Copenhagen University Hospital), Copenhagen, Denmark
- France (9):
  - CHU de Besancon, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - Hôpital Cochin, Paris
  - CHU Poitiers - Hôpital la Milétrie, Poitiers
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Italy (2):
  - IEO Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Med-Polonia Sp. z o.o, Poznan, Poland
- Spain (9):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Ruber Internacional, Madrid
  - Centro Oncologico Clara Campal, Madrid
  - Hospital Universitary Fundacion Jimenez Diaz, Madrid
  - NEXT Oncology Madrid, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (3):
  - St Bartholomews Hospital, London
  - University College London Hospital, London
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No